CLINICAL TRIAL: NCT01517516
Title: A Magnetic Resonance Imaging (MRI) Study to Investigate Differences in the Structure and the Function of the Brain at Rest; Between Persons With Functional Pain Conditions Such as IBS or Vulvodynia, IBD and Healthy Controls
Brief Title: Multi Modal Imaging: An MRI Study to Investigate Differences in the Structure and the Function of the Brain at Rest.
Acronym: MMI
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emeran Mayer, MD, Professor, Department of Medicine at the David Geffen School of Medicine, UCLA, University of California, Los Angeles
Other Study IDs: 11-000069; RO1 DKO48351 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2011-12-14; First posted 2012-01-25 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome; Cyclical Vomiting Syndrome; Ulcerative Colitis; Vulvodynia; Crohn's Disease
Keywords: fMRI; resting state; structural MRI; functional MRI
MeSH Terms: conditions — Irritable Bowel Syndrome; Familial cyclic vomiting syndrome; Colitis, Ulcerative; Vulvodynia; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Functional Pain Conditions and Inflammatory bowel disease: Cyclical Vomiting Syndrome, Irritable Bowel Syndrome, Inflammatory Bowel disease (Ulcerative colitis and Crohns)and Vulvodynia (vestibulodynia)
- Inflammatory Bowel Disease: Subjects diagnosed with Crohn's Disease or Ulcerative Colitis.

SUMMARY:
The structural/RSN study involves Structural and Resting State Neuroimaging. The purpose of Structural Neuroimaging is to use MRI technology to identify cortical and white matter morphometric differences between patients with chronic pain conditions and healthy control subjects.

The purpose of the Resting State Neuroimaging study is to use functional MRI to identify possible disease related differences in various resting state networks in the brain.

In addition we are looking at the effect gut microbiota on brain function in healthy and IBS participants.

The overall goal is to identify structural and functional brain differences in persons with chronic pain conditions such as Irritable Bowel Syndrome (IBS, Cyclical Vomiting Syndrome(CVS) and vestibulodynia/vulvodynia. We are also looking at Inflammatory Bowel Disease(ulcerative colitis and Crohn's disease. We will be comparing differences between these conditions and matched healthy control subjects.

DETAILED DESCRIPTION:
The study involves 2 visits. The screening visit is about 90 minutes and involves signing the consent, completing questionnaires, a medical history, modified physical exam and psychological interview to identify stressors, anxiety, depression and other conditions.

The second visit is the MRI visit (both functional and structural) and also will take about 90 minutes, with the scanning lasting about 45 minutes. There are questionnaires and a measure of skin conductance also.

We have added a single stool sample for microbiota analysis and a food frequency questionnaire in the healthy control and IBS populations.

ELIGIBILITY:
Inclusion Criteria:

Men and women who meet the following criteria are eligible for inclusion in the study:

1. 18 to 55 years of age
2. ROME III criteria for IBS population
3. Willingness to participate in this study as evidenced by a signed, written informed consent form (ICF).
4. If female and of childbearing potential willingness to avoid pregnancy and practice adequate birth control (abstinence, oral contraception, intrauterine devices, implantable devices, depot contraceptives, or barrier method with spermicide) during the time of study enrollment.
5. If female, negative urine pregnancy tests at Screening Visit 1, and visit 2.
6. Right handed
7. Ambulatory outpatient (not depending exclusively on a wheelchair for mobility)
8. English is primary oral and written language.
9. Diagnosed with CVS
10. Diagnosed with IBD and currently not taking steroid therapy.
11. Diagnosed with vestibulodynia (a subgroup of vulvodynia)
12. Pre and peri menopausal only, post menopausal excluded.

Exclusion Criteria:

1. Evidence of structural abnormality of the gastrointestinal tract. Subjects with Functional GI conditions must be without 'red flags', that may indicate gastrointestinal disease. Exclusionary GI conditions include but are not limited to: gastrointestinal surgery (exceptions: IBD group, appendectomy, benign polypectomy, cholecystectomy)also esophagitis, celiac disease, gastrointestinal malignancy or obstruction; peptic, duodenal or gastric ulcer disease.
2. Clinical evidence of cardiovascular, respiratory, renal, hepatic, malignancy, hematologic, neurologic, psychiatric or any disease that the PI determines may interfere with safe participation in the study
3. Use of investigational drugs, products or devices within 28 days prior to screen and through study participation.
4. Subjects with current regular use of narcotics and or opioids. Use of medications/drugs that affect the central nervous system. TCA's, SSRI's or other antidepressants are allowed if on stable dose for 3 months or more.
5. Pregnancy or breast feeding
6. Subjects with extreme obesity (BMI > 35%)
7. Subjects with metal implants, dental retainers, large tattoos (e.g. full arm or back) or claustrophobia; making MRI safety not possible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from clinics, community in and around Los Angeles Area.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Resting state networks | within 1 week of scanning visit
  The resting state functional MRI scan will be done to assess differences in the resting state networks in subjects with chronic pain conditions in comparison to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Emeran Mayer, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Gail and Gerald Oppenheimer Family Center for Neurobiology of Stress, Los Angeles, California, United States